CLINICAL TRIAL: NCT02766686
Title: Preference-based Comparative Study on Definitive Radiotherapy of Prostate Cancer With Protons in Standard Fractionation and Standard Dosage
Brief Title: Preference-based Comparative Study on Definitive Radiotherapy of Prostate Cancer With Protons
Acronym: ProtoChoice-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Consortium for Translational Cancer Research (Other); National Center for Radiation Research in Oncology Dresden/Heidelberg (Other); Radiation Oncology Working Group of the German Cancer Society (Other)
Responsible Party: Principal Investigator, Tobias Hölscher, Dr. Tobias Hölscher, Technische Universität Dresden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR - ProtoChoice-P - 2015
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; proton radiotherapy; photon radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Protons; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiotherapy with protons (Experimental): Proton radiotherapy 74-80 Gray equivalent (GyE), 2Gy per fraction, 5 fractions peer week
  Interventions: Radiation: Radiotherapy with protons
- Radiotherapy with photons (Active Comparator): Photon-Intensity-Modulated Radiation Therapy (IMRT) without lymph drainage vessels, 74-80 Gy, 2Gray (Gy) per fraction, 5 fractions peer week
  Interventions: Radiation: Radiotherapy with photons
- Radiotherapy with photons with lymph drainage vessels (Other): Photon-IMRT with lymph drainage vessels, 74-80 Gy, 2Gy per fraction, 5 fractions peer week
  Interventions: Radiation: Radiotherapy with photons

INTERVENTIONS:
Radiation: Radiotherapy with protons
  Arms: Radiotherapy with protons
Radiation: Radiotherapy with photons
  Arms: Radiotherapy with photons; Radiotherapy with photons with lymph drainage vessels

SUMMARY:
ProtoChoice-P is a prospective multicenter trial to evaluate proton therapy in patients suffering from prostate cancer. Primary aim of the study is a decrease of moderate or severe genito-urinary or intestinal side effects (Common Terminology Criteria for Adverse Events (CTCAE) 4.0 grade 2 or higher) by the use of proton therapy. Secondary endpoints contain assessment of quality of life, biochemical recurrence and recurrence free survival as well as overall survival and economic comparison between photon and proton therapy.

DETAILED DESCRIPTION:
The hypothesis of the study is a 7.5% decrease of combined genito-urinary and intestinal side effects from 15% with photon therapy to 7.5% by the use of protons. With an alpha of 0.05 and 80% power it is therefore necessary to treat 131 patients with protons to detect such difference. With an estimated drop-out rate of 10% 146 patients have to be recruited to the proton arm. As randomization to photon or proton therapy is not possible in a multicenter setting with only few proton facilities available patients treated with photons will be prospectively matched to their proton counterparts. Stratification criteria will include: Age, high dose volume, androgen deprivation, history of surgery, obstructive disease, increased risk for rectal bleeding, socio-economic criteria and use of rectal balloon during radiotherapy. Comparison of the primary endpoint will be restricted to patients without irradiation of lymphatic drainage.

ELIGIBILITY:
Inclusion Criteria:

* life expectancy ≥ 10 years
* adenocarcinoma of the prostate confirmed by punch biopsy
* locally limited to locally advanced adenocarcinomas without evidence of distant metastases i.e. T1-3b N0-1 M0
* stage-related indicated neoadjuvant / adjuvant androgen deprivation possible (neoadjuvant ≤ 6 months)
* good general condition (ECOG performance status 0 - 1)
* marker seed implantation before irradiation (optional) or possibility of Image-guided Radiation Therapy (IGRT) by CT
* adequate compliance for follow-up
* written informed consent

Exclusion Criteria:

* distant metastases
* previous radiotherapy of the lesser pelvis
* previous or concomitant other malignant disease except when there is no impact on treatment or follow-up of the prostate cancer
* participation in another clinical study, if it's excluded by the study protocols

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of moderate/ severe side effects | after 2 years ( measured from the first day of treatment)
  ≥ grade 2 by CTCAE combined for genito-urinary and gastrointestinal side effects

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hölscher, Dr., Study Chair — University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, German Consortium for Translational Cancer Research (DKTK)
Locations (3):
- Germany (3):
  - University Hospital Carl Gustav Carus, Department of Radiotherapy and Radiation Oncology, Dresden
  - Klinikum rechts der Isar, Technische Universität München, Munich
  - Universitätsklinik für Radioonkologie, Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No